CLINICAL TRIAL: NCT01483339
Title: Metacognitive Therapy Versus Exposition With Response Prevention for Patients With Obsessive-Compulsive Disorder
Brief Title: Metacognitive Therapy for Patients With Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Psychotherapie-Ambulanz Marburg e.V. (Other)
Responsible Party: Principal Investigator, Julia Anna Glombiewski, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT_OCD_2011
Record Dates: First submitted 2011-11-16; First posted 2011-12-01 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metacognitive Therapy (Experimental)
  Interventions: Behavioral: Metacognitive Therapy
- Exposure and Response Prevention (Experimental)
  Interventions: Behavioral: Exposure and Response Prevention

INTERVENTIONS:
Behavioral: Metacognitive Therapy — Metacognitive Therapy for OCD according to Wells (1997)
  Arms: Metacognitive Therapy
Behavioral: Exposure and Response Prevention — Exposure and Response Prevention for OCD according to Kozak & Foa (1997)
  Arms: Exposure and Response Prevention

SUMMARY:
Cognitive behavior therapy is the most effective treatment of obsessive-compulsive disorder. However, the majority of treated patients remain symptomatic. The metacognitive therapy by Wells (1997) could achieve substantial gains in first pilot studies. The purpose of this study is to investigate this approach with a randomized controlled trial by comparing metacognitive therapy with exposure and response prevention for obsessive-compulsive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: obsessive-compulsive disorder
* German-speaking
* Agreeing to participate, verified by completion of informed consent

Exclusion Criteria:

* Current or past diagnosis of substance dependence, psychosis, neurological conditions
* Mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity (Yale Brown Obsessive-Compulsive Scale; YBOCS) from Pretest to Posttest to Follow-up | from Pretest (admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)

SECONDARY OUTCOMES:
Change in Symptom Severity (Padua Inventory; PI) from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to two in-between timepoints (an expected average of 5 and 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
Change in Metacognitions from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to two in-between timepoints (an expected average of 5 and 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  Metacognitions (MCQ), Thought Fusion Inventory (TFI), Thought Action Fusion Scale (TAF-scale), Beliefs About Rituals Inventory (BARI), Stop Signals Questionnaire (SSQ), Detached Mindfulness Questionnaire (DMQ)
Change in Obsessive Beliefs (Obsessive-Beliefs Questionnaire, OBQ) from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to two in-between timepoints (an expected average of 5 and 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
Change in Behavioral Avoidance (Behavioral Avoidance Test, BAT) from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to two in-between timepoints (an expected average of 5 and 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
Change in Depression (Beck Depression Inventory, BDI) from Pretest to Posttest to Follow-up | from Pretest (admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
Change in Anxiety (Beck Anxiety Inventory, BAI) from Pretest to Posttest to Follow-up | from Pretest (admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
Change in Patient-Therapist-Alliance from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to two in-between timepoints (an expected average of 5 and 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
  Self rating and clinician rating of Helping Alliance Questionaire (HAQ) and Working Alliance Inventory (WAI)
Change in Symptom Severity (Clinical Global Impressions; CGI) from Pretest to two in-between timepoints to Posttest to Follow-up | from Pretest (admission) to two in-between timepoints (an expected average of 5 and 10 weeks after admission) to Posttest (an expected average of 3 months after admission) to Follow-up (an expected average of 6 months after admission)
Treatment expectancy (Treatment Expectancy Questionnaire) after the first treatment session | after the first treatment session (an expected average of 1 week after admission)
Satisfaction with the treatment at Posttest | immediately after completion of therapy (an expected average of 3 months after admission)
Change in Symptom Severity (Obsessive-Compulsive Disorder Scale; OCD-S) measured before every treatment session | from the first treatment session (an expected average of 1 week after admission) to the last treatment session (an expected average of 3 months after admission) on a weekly basis

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Exner, Prof. Dr., Principal Investigator — University of Leipzig; Winfried Rief, Prof. Dr., Study Director — Philipps University Marburg, Department of Clinical Psychology and Psychotherapy
Locations (1):
- Philipps Univerity Marburg, Department of Clinical Psychology and Psychotherapy, Marburg, Hesse, Germany

REFERENCES:
- See also: Related Info — http://www.uni-marburg.de/fb04/ag-klin/pam